# Implementing the MSK-HQ to empower patients and improve services

# The MSK-Tracker study

18/12/2018

# **RESEARCH REFERENCE NUMBERS**

IRAS Number: 237571

ISRCTN / Clinical trials.gov Number: RG-0132-16-IPCHS

**Sponsor Number:** RG-0132-16-IPCHS

**Funder's Number:** 21405 (Arthritis Research UK)

# **KEELE STATISTICAL ANALYSIS PLAN (SAP)**

Title: The MSK Tracker single centre before & after sequential comparison study.

# Study team:

Dr Jonathan Hill, Steven Blackburn, Georgina Craig, Krysia Dziedzic, Steff Garvin, Elizabeth Gibbons, Elaine Hay, Gillian Lancaster, Gareth McCray, Ajit Menon, Andrew Price, Joanne Protheroe, Kay Stevenson, Katie Tempest, and Steph Tooth.

#### Authors of the SAP:

| Draft numberversion 1.4 | Date05/12/2018 |
|--------------------------------------|------------------|
| Chief InvestigatorJonathan Hill | Signature (Date) |
| Principal InvestigatorJonathan Hill | Signature (Date) |
| Study Statistician Gareth McCray | Signature (Date) |
| Senior StatisticianGillian Lancaster | Signature (Date) |

#### Declaration regarding undertaking of the analysis

Gareth McCray will be undertaking data cleaning and analysis of the study data under the guidance and supervision of Gillian Lancaster.

#### With reference to Protocol version ...1.0 06 March 2018.

# **Version History Log**

This section should detail the key elements of the changes to the successive versions.

| Version | Date<br>implemented | Section no.<br>changed | Details of changes |
|---|---|---|---|
| 1.1 | 25/05/2018 | Up to section<br>5 | Jonathan made some minor changes that were suggested by Gillian Lancaster |
| 1.2 | 27/07/18 | Sections 5-7,<br>9 | Gareth updated sections 5-7, 9,10 |
| 1.3 | 18/09/18 | As above | Gill made some edits to text and tables |
| 1.4 | 05/12/2018 | All | Gareth made edits to final tables and text |

# **Contents page**

| | Page No |
|-----------------------------------------|---------|
| 1 Background and Aims | 4 |
| 2 Design | 4 |
| 3 Study population | 5 |
| 4 Outcomes | 5 |
| 5 Sample size | 6 |
| 6 Population (baseline) characteristics | 6 |
| 7 Methods of analysis | 7 |
| 8 References | 8 |
| 9 Tables | 9 |
| 10 Appendix | 17 |

# Glossary of terms / Abbreviations (list) ...

BMJ British Medical Journal

BOA British Orthopaedic Association

CATS Clinical Assessment and Treatment Services

CI Chief Investigator

CRF Case Report Form

CSP Chartered Society of Physiotherapy

CTU Clinical Trials Unit

DoH Department of Health

EBCD Experience Based Co-Design

ELC Experience Led Commissioning

e-PROM electronic - Patient Reported Outcome Measure

GCP Good Clinical Practice

GDPR General Data Protection Regulation

HRA Health Research Authority

ISRCTN Trials Number International Standard Randomised Controlled

MSK Musculosketal

MSK-HQ Musculoskeletal Health Questionnaire

NICE National Institute for Health and Care Excellence

NHS National Health Service
PI Principal Investigator

PPIE Patient & Public Involvement & Engagement

PROM Patient Reported Outcome Measure

QI Quality Improvement

QiPP programme Quality, Innovation, Productivity and Prevention

RCGP Royal College of General Practitioners

RUG Research User Group
SAE Serious Adverse Event

SFTP Secure File Transfer Protocol
SOP Standard Operating Procedure

SSL Secure Sockets Layer

#### 1. Background and Aims

The Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) is a recently validated new MSK Patient Reported Outcome Measure (PROM) that has been co-produced with patients and clinicians to measure the holistic impact of an MSK condition on a person's health. However, it is not yet known whether:

- Patients using the MSK-HQ routinely as part of their care planning, supports them to feel more involved and empowered in managing their health issues.
- Using the MSK-HQ can facilitate a more holistic care planning consultation, both in terms of the quality of patient interactions and communications with healthcare professionals.
- It is acceptable or feasible for both patients and clinicians to use the MSK-HQ as an e-PROM.

Enabling organisations to examine their aggregated MSK-HQ data at service level may also help to identify unmet need, improvement opportunities and inform MSK service and organisational developments.

The overall aim of this research is to co-design and test the feasibility and impact of implementing the MSK-HQ presented within an innovative online care planning package called the MSK-Tracker. Secondary objectives are:

- a) To optimise the acceptability and utility of the MSK-Tracker as a self-management support tool for patients to use to take control of their MSK health issues and facilitate personal goal setting during MSK clinical encounters
- b) To assess the feasibility and utility of the MSK-Tracker in busy consultations; the impact on the nature of the consultation when the MSK-Tracker is used and whether it supports patient enablement (feeling more in control of their MSK condition).
- c) To assess its value in generating aggregated outputs and insight to inform service improvement and organisational development of MSK interface services.

#### 2. Design

The study is using a 'before' and 'after' sequential comparison design with an iterative pilot and user testing phase in between. In addition, audio recordings of the consultation (in a sub-sample, n=40 (phase 1=20 & phase 3=20)), alongside individual clinician (n=10) and patient interviews and a feedback workshop with clinicians and patients, will explore the feasibility, and impact of implementing the MSK-Tracker within routine consultations and user experiences. The study will take place in Staffordshire Musculoskeletal Interface Service based at Haywood Hospital in Burslem, Stoke-on-Trent.

# 3. Study and evaluative population

Patients aged 18 years and above with an appointment to attend the Staffordshire Musculoskeletal Interface Service for an MSK pain problem will be invited to take part. Patients unable to use or access the internet will be unable to take part in this research as well as patients who do not provide informed consent for study participation and data collection. The online system will only be available in English.

**Phase 1 ('Before' stage).** Patients (n=120) who meet the eligibility criteria for having long-term MSK pain will consent online and complete an electronic survey shortly before their consultation. This phase will not utilise the new innovative 'MSK-Tracker' online components, in order to give a baseline comparator. Patients will complete follow-up data 2 weeks and 3 months after their clinic date and clinicians will complete a case report form (CRF) using the clinician portal. Audio recordings of approximately 20 patient consultations will examine consultation conversations and their content using discourse analysis.

**Phase 2. ('Pilot stage').** Phase 2 will focus on pilot testing the MSK-Tracker components including the, pre-clinic preparation survey, clinician dashboard, summary action plan, patient's goal setting module, follow-up survey and progress charts. The study will seek to refine the processes used in phase 3, with a limited number of patients (approximately 40 patients in 2 cycles of 20) and clinicians (n=10) using the Tracker.

Phase 3 ('After' stage). Stage 3 will mirror Phase 1, with newly recruited patients, except the final MSK-Tracker components will be used. As in phase 1, audio recordings of approximately 20 patient consultations will examine consultation conversations and their content. In addition, a report will be produced for the clinical managers about their service outcomes and areas of unmet need in order to inform quality improvement with a workshop planned to better understand what information services find most useful.

#### 4. Outcomes

For each of the study Phases (1-3), taken at Baseline, Two-week follow-up and/or three month follow up (see section 9 for details on the specific measures collected at each time point).

#### Baseline measures:

 A range of patient self-report characteristics to be able to describe the patient population such as age, gender, ethnicity, education level, work status, health literacy, MSK pain site/condition, and episode duration. See Tables in section 9 of this document.

#### Primary outcome measure:

The Patient Enablement Index (PEI)

#### Secondary outcome measures:

 A number of secondary outcomes will be collected including: MSK-HQ score, Consumer Health Activation Index score, consultation experience measures, work status and impressions of the MSK-tracker system. See Tables in section 9 for full details of these outcomes and how they will be reported.

#### Feasibility outcomes:

A range of feasibility outcomes will be reported, including: numbers of participants
completing each stage of the study, details around study registration, 2-week followup and 3-month follow-up, timing of and time taken to complete study survey
components. See Tables section 9 for full details of what feasibility information will
be collected and how it will be reported.

#### 5. Sample size

The primary outcome of this trial is the patient enablement instrument (PEI)¹ at 2 week follow up. As patients are asked to retrospectively rate the level of enablement, at the 2-week follow up, as a result of their visit to the Staffordshire Musculoskeletal Interface Service we only have a score at a single time point (and not a change score) for each group of patients in Phase 1 and Phase 3. The Patient Enablement Instrument consists of six items graded on three-point scales. It is scored between 0 and 12 and a high score represents more enablement. The sample size was generated based on that required for an independent groups two-sample t-test with a two tailed 5% significance level at 80% power. As no Minimally Clinically Important Difference (MCID) relevant to the specific context could be found for the PEI, the study is powered to find a 0.40 effect size — representative of a small to medium effect.² The expected SD for the population is 3.86¹ (taken from Howie et al. 1998) thus, the implied MCID between the groups would be a score of 1.55 scale points. Accordingly, the required sample is 100 in each arm. If we account for 20% dropout and missingness, the target recruitment is 120 in both phases 1 and 3.

#### 6. Participant characteristics

Baseline characteristics for participants will be displayed in relation to the two groups of participants, i.e., those who are enrolled Phase 1 and those who are enrolled in Phase 3. Given the fact that patient groups are not randomly allocated hypothesis testing will be done comparing the groups at baseline for comparability.

**See Tables in section 9** for details of which variables will be collected and how they will be reported.

#### 7. Methods of analysis

#### **Descriptive statistics:**

For all outcomes, numerical variables will be summarised as either mean (SD) or median (IQR) depending on the skew of the distribution of the variable in question. Categorical variables will be described as frequencies and percentages.

#### Primary outcome measure:

A two-tailed independent sample t-test will be conducted to compare the mean PEI score in Phase 1 with that in Phase 3. An effect size, Cohen's Delta, and 95% confidence intervals will be reported for the mean difference between scores. A p-value will be reported with a significance level rate of < 5% leading to a rejection of the null hypothesis of no difference between the two groups.

Model residuals will be checked for normality, if deviation is found appropriate transformations will be made to the PEI score. Exploration of patterns of missingness will be undertaken to look for potential associates with baseline. Under the assumption of Missing at Random (MAR) missing data on the primary outcome measure will be imputed via the multiple imputation by chained equation (MICE) method<sup>3</sup>. Sensitivity analysis will be conducted to assess impact of the MAR assumption. Analyses will be done with missing values both  $\pm 1.55$  scale points (the implied MCID) on the PEI – to model the potential effect of Missing Not at Random Bias (truncated between 0 – 12).

#### Secondary outcome measures:

Secondary outcome measures will be analysed via t-test. Effect sizes and 95% confidence intervals will be reported for all measures. P-values will be reported and a <5% rejection criterion will be utilised. No sensitivity analyses will be undertaken and no corrections for multiplicity will be made for the secondary outcomes.

#### Feasibility outcomes:

Only descriptive statistics for the feasibility outcomes will be reported. These will be counts and percentages with an appropriate denominator for each measure.

#### **Technical details:**

It is envisioned that R (current version 3.5.1) will be used for all analyses. The primary outcome will be analysed by the two study statisticians, unblinded. The statistical analyses and associated datasets will be kept in the appropriate section of the trial master file on the internal secure network.

#### 8. References

1. Howie JG, Heaney DJ, Maxwell M, Walker JJ. A comparison of a patient enablement instrument (PEI) against two established satisfaction scales as an outcome measure of

- primary care consultations. Fam Pract. 1998;15(2):165-171.
- 2. Cohen J. A Power Primer. *Psychol Bull*. 1992;112(1):155-159.
- 3. Buuren S, Groothuis-Oudshoorn K. mice: Multivariate imputation by chained equations in R. *J Stat Softw.* 2011;45(3).

# 9. Tables/Figures

Feasibility/process outcomes

| Potential participants | Phase 1 (before) | Phase 3 (after) | Total |
|---|---|---|---|
| Number of patients invited to take part | | | |
| Actual participants: | | | |
| Study consent & Completed baseline survey | | | |
| Consultation audio recording | | | |
| Clinician completed case report form in clinic | | | |
| Patient received clinic summary action plan | | | |
| Accessed goal setting module | | | |
| Patient completed 2-week FU survey | | | |
| Patient needed a reminder email for 2-week FU survey | | | |
| Patient completed 3-month FU survey | | | |
| Patient needed a reminder email for 3-month FU survey | | | |
| Timing of survey completion: | | | |
| Time from completion of baseline survey to clinic – Mean (SD), days | | | |
| Time from clinic to 2-week FU survey completion – Mean (SD), days | | | |
| Time from clinic to 3-month FU survey completion – Mean (SD), days | | | |
| Time take to complete survey: | | | |
| Baseline survey – Mean (SD), mins* | | | |
| 2-week FU survey – Mean (SD), mins* | | | |
| 3-month FU survey – Mean (SD), mins* | | | |

#### Baseline characteristics at Phase 1 and Phase 3

| Characteristic | Phase 1 (before) | Phase 3 (after) | Total | Mean (95% CI) | P-value |
|---|---|---|---|---|---|
| Demographics | | | | | |
| Age - Mean (SD) | | | | | |
| Sex: | | | | | |
| Male | | | | | |
| Female | | | + | | |
| Prefer not to say | | | | | |
| Missing | | | | | |
| Ethnicity: | | | | | |
| Mixed | | | | | |
| Asian | | | | | |
| Black | | | | | |
| White | | | | | |
| Other | | | | | |
| Prefer not to say | | | | | |
| Missing | | | | | |
| Problem Characteristics | | | | | |
| Pain Location(s) (percentage of respondents overall): | | | | | |
| Head region | | | | | |
| Neck | | | + | | |
| Shoulder/upper arm | | | | | |
| Lower arm/wrist | | | + | | |
| Hand(s) | | | | | |
| Upper back/chest/abdomen | | | | | |
| Lower back/pelvis | | | | | |
| Hip, groin, thigh | | | | | |
| Knee/lower leg | | | | | |
| Ankle/foot | | | | | |
| Other | | | | | |
| (percentage of respondents overall) | | | | | |
| Single site pain | | | | | |
| Multiple sites pain (more than one pain location) | | | | | |
| Has diagnosis – No. (%) | | | | | |
| Missing | | | | | |
| Problem duration: | | | | | |
| < 2 weeks | | | | | |
| 2 to 4 weeks | | 1 | + | | |
| 5 weeks to 3 months | | | + | | |
| 4 to 6 months | | | <del> </del> | | |
| | | | 1 | | |
| 7 to 12 months | | | 1 | | |
| 13 months to 3 years | | | | | |
| > 3 years | | | | | |
| Missing | | | 1 | | |
| Previous physio for problem –No. (%) | | | | | |
| Missing | | | | | |
| Previous surgery for problem: | | | | | |
| No related surgery | | | | | |
| 1 related surgery | | | | | |
| 2 related surgeries | | | 1 | | |
| 3 or more related surgeries | | | + | | |

| | | ı | 1 |
|---|---|---|---|
| Missing | | | |
| Referral source: | | | |
| GP | | | |
| Self-referral | | | |
| Orthopaedic Surgeon | | | |
| Neurologist/Neurosurgeon | | | |
| Occupational Health | | | |
| Other | | | |
| Missing | | | |
| Medication usage for problem | | | |
| Missing | | | |
| Comorbidities: | | | |
| Heart disease | | | |
| High blood pressure | | | |
| Poor circulation | | | |
| Lung disease | | | |
| Diabetes | | | |
| Kidney disease | | | |
| Neurological disorder (e.g. stroke) | | | |
| Liver disease | | | |
| Cancer | | | |
| Depression | | | |
| Arthritis | | | |
| None | | | |
| Number of Comorbidities – Mean(SD) | | | |
| Independence: | | | |
| Needed assistance to fill in this questionnaire | | | |
| Considers self to have a carer | | | |
| Health Literacy | | | |
| Help needed to read instructions on pamphlets or other written | | | |
| material from your doctor or pharmacy – ("often" or "always") (%) | | | |
| Work & Activity | | | |
| <del>-</del> | | | |
| Work status – Working | | | |
| Missing | | | |
| Hours missed from work in last 7 days because of problem- Mean | | | |
| (SD) (only working patients) | | | |
| Hours missed from work in last 7 days for other reasons- Mean (SD) | | | |
| (only working patients) | | | |
| Hours worked in last 7 days - Mean (SD) (only working patients) | | | |
| Joint and muscle symptoms affect your productivity while working - | | | |
| Mean (SD) (only working patients) | | | |
| Joint and muscle symptoms affect ability to do regular daily | | | |
| activities, other than work - Mean (SD) (only working patients) | | | |
| WPAI Derived Measures: | | | |
| Percent work time missed due to problem: | | | |
| Percent impairment while working due to problem | | | |
| Percent overall work impairment due to problem | | | |
| Percent activity impairment due to problem | 1 | | |

#### Outcome measures at baseline:

| Overall MSK Health Status |
|---|
| MSK-HQ score – Mean (SD) |
| [score range goes from 0 – 56: higher score are milder symptoms] |
| Reference values: |
| <ul> <li>Mean MSK-HQ in National FCP pilot = 34</li> </ul> |
| <ul> <li>Mean MSK-HQ in Community physio = 32</li> </ul> |
| <ul> <li>Mean MSK-HQ in GP sample = 30</li> </ul> |
| <ul> <li>Mean MSK-HQ in Ortho hip and knee waiting list sample = 27</li> </ul> |
| Patient Activation Level |
| The Consumer Health Activation Index (CHAI) score – Mean (SD) |
| [score range goes from 0-100: higher score is greater health |
| engagement, understanding, confidence and knowledge] |
| Reference values: |
| <ul> <li>In a sample of 10,000 American adults, mean CHAI was 80.</li> </ul> |
| Low (CHAI score 0-79) |
| Moderate (CHAI score 80-94 |
| High (CHAI score 95-100) |

Conclusion: There were no differences in patient outcomes between before and after phases

Case Report form completed by clinicians online

| case Report form completed by clinicians offine | | | |
|-------------------------------------------------|---------|---------|-------|
| | Phase 1 | Phase 3 | Total |
| | (n=93) | (n=83) | |
| Review Decision | | | |
| Review | | | |
| ReviewPendingResults | | | |
| SOS Appt | | | |
| Discharged | | | |
| Treatment decision | | | |

| | 1 | I |
|---|---|---|
| Injection Given | | |
| Injection Given Opt (IM) | | |
| Injection Given Opt (SC) | | |
| Injection Given Opt (IA) | | |
| Advice Given | | |
| Treatment Declined | | |
| No Change To Current Treatment | | |
| No Treatment Needed | | |
| Treatment Recommendations To GP | | |
| New Treatment Started | | |
| Amendments To Current Treatment | | |
| Investigations | | |
| Immunology | | |
| Microbiology | | |
| Xray | | |
| MRI | | |
| MRIOpt | | |
| USound | | |
| CTScan | | |
| SynovialFluid | | |
| Isotope | | |
| Echo | | |
| ECG | | |
| PFT | | |
| Haematology | | |
| Biochemistry | | |
| MSSU | | |
| 24HrUrine | | |
| Capillaroscopy | | |
| Dexa | | |
| Neurophysiology | | |
| Other | | <br> |
| Referrals | | |
| Physio | | |
| Podiatry | | |
| OT | | |
| Splinting | | |
| Orthotics | | |
| Chronic Pain | | |
| Chronic rain | | |
| Pain Clinic | | |
| Pain Clinic | | |
| Clinical Diagnoses: | | |
| Clinical Diagnoses:<br>Shoulder | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elibow Epicondylitis Olecranon Bursitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis Rodes OA | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis ACA Other | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis AOA Other Hip | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Copal | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis OA Other Hip | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis AOA Other Hip Other Hip Other Piriformis Meralgia Paraesthetica | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCIOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis Acado Other Hip Other Hip Other Hip Other Piriformis Meralgia Paraesthetica Adductor Enthesopathy | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCJOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis OA Other Hip Other Hip Other Piriformis Meralgia Paraesthetica Adductor Enthesopathy Ischiogluteal Bursitis | | |
| Clinical Diagnoses: Shoulder Adhesive Capsultis GlenohumeralOA ACJOA Subacromial Bursitis Rotor Cuff Impingement Calcific Tendomitis Rotator Cuff Tear Bicipital Tendonitis Rotator Cuff Tear Type Crystal Arthropathy Instability Other Hand / Wrist Trigger Finger First CMCIOA No dalOA De Quervains Tenosynovitis Ganglions Carpal Tunnel Syndrome Ulnar Neuritis Radiocarpal OA Other Elbow Epicondylitis Olecranon Bursitis Loose Body Ulnar Neuritis Acado Other Hip Other Hip Other Hip Other Piriformis Meralgia Paraesthetica Adductor Enthesopathy | | |

| 04 | I |
|---|---|
| OA OA | |
| Spine | |
| Other | |
| Coccydinia | |
| Osteoporotic Vertebral Fracture | |
| Spinal Stenosis | |
| Serious Spinal Pathology | |
| Chronic Low Back Pain | |
| Back Pain With Nerve Root Pain | |
| Low Back Pain | |
| Knee | |
| Other | |
| Shin Splints | |
| Pseudogout | |
| Pyrophosphate | |
| Cruciate Ligament Injury | |
| Collateral Ligament Injury | |
| Tendonitis | |
| Bursitis | |
| Bakers Cyst | |
| Anterior Knee Pain | |
| Menisceal Tear | |
| Mensical Degeneration | |
| Pateliofemoral OA | |
| Tibiofemoral OA | |
| Foot / Ankle | |
| Pain Arthritis | |
| Ligamentous Injury | |
| Instability | |
| Achilles Rupture | |
| Achilles Tendiopathy | |
| Tendinitis | |
| Subtelar Joint Arthritis | |
| Pes Planual | |
| Mid Foot Pain OA | |
| Mortons Neuroma | |
| Metatarsalgia | |
| Hallux Valgus | |
| First MTPJOA | |
| Plantar Fascitis | |
| Gout | |
| Other | |
| Neck | |
| Cervical Spondylosis | |
| Cervical Spondylosis<br>Mechanical Neck Pain | |
| Cervical Spondylosis<br>Mechanical Neck Pain<br>Brachial Neuritis | |
| Cervical Spondylosis<br>Mechanical Neck Pain<br>Brachial Neuritis<br>Radiculopathy | |
| Cervical Spondylosis<br>Mechanical Neck Pain<br>Brachial Neuritis<br>Radiculopathy<br>Non Specific Neck Pain | |
| Cervical Spondylosis<br>Mechanical Neck Pain<br>Brachial Neuritis<br>Radiculopathy<br>Non Specific Neck Pain<br>Other | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Polymyalgia Malignancy Other Refer | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy Other Refer | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Hoffer Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Ortho For Opinion Other Other Clinical diagnosis | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Halignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Opther Other Clinical diagnosis | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Alignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other For Opinion Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Halignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Hypermobility Polymyalgia Other Refer Combined Clinic Ortho For Opinion Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: | |
| Cervical Spondylosis Mechanical Neck Pain Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Hydrotherapy | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Malignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Hydrotherapy Splint Orthotics | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Halignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Hydrotherapy Splint Orthotics | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Adlignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Required during admission: Poditry Spelific Orthotics Poditry Specific | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Halignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Hydrotherapy Splint Orthotics | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Halignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Reditry Spelific Poditry Spelific | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Halignancy Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Repolitry Splint Orthotics Poditry Specific Poditry Specific | |
| Cervical Spondylosis Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Hypermobility Other Refer Combined Clinic Orthopaedics For Surgery Pending Results Refer To Ortho Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Hydrotherapy Splint Orthotics Specific Other Other Other Other Other Other Other Orthopaedics For Surgery Pending Results Refer To Ortho Other Other Other Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: OT Physio Poditry Splint Orthotics Specific | |
| Cervical Spondylosis Mechanical Neck Pain Mechanical Neck Pain Brachial Neuritis Radiculopathy Non Specific Neck Pain Other Other Diagnosis Fibromyalgia Inflammatory Arthritis Chronic Widespread Pain Gout Hypermobility Polymyalgia Hypermobility Polymyalgia Other Refer Combined Clinic Ortho For Opinion Other Other Clinical diagnosis Copy GP Letter To Patient Included In Research Trials And Education No Notes For Patient In Clinic Required during admission: Required during admission: Genticula Specific Other Othopadics For Surgery Pending Results Refer To Orthopadics For Surg | |

Two week follow up on outcome measures

| | Phase 1 | Phase 3 | Total | Mean (95% CI) | P-value |
|---|---|---|---|---|---|
| Global change in MSK condition since my clinic appointment | | | | <u> </u> | |
| (5 =much better to 1 = much worse- see below) – Mean (SD) | | | | | |
| Global change | | | | | |
| 5. Much better | | | | | |
| 4. Better | | | | | |
| 3. Same | | | | | |
| 2. Worse | | | | | |
| 1. Much worse | | | | | |
| Composite Scores | | | | | |
| Patient enablement index – Mean (SD) | | | | | |
| [score range is 0 to 12: higher scores = better empowerment] | | | | | |
| This items asks – "As a result of your visit to the clinic, do you | | | | | |
| feel you are:" (options - Much better=2, Better=1, Same=0) | | | | | |
| Able to understand your illness | | | | | |
| Able to cope with your illness | | | | | |
| <ul> <li>Able to keep yourself healthy</li> <li>Able to cope with life</li> </ul> | | | | | |
| Confident about your health | | | | | |
| Able to help yourself | | | | | |
| Reference values: | | | | | |
| In a GP sample patient mean PEI score was 4 points (1 wk later) | | | | | |
| MSK-HQ score – Mean (SD) | | | | | |
| , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | | | | |
| Reference score at Follow-up: | | | | | |
| Mean MSK-HQ in National FCP pilot = 41 | | | | | |
| <ul> <li>Mean MSK-HQ in Community physio = 42</li> </ul> | | | | | |
| Mean MSK-HQ in GP sample = 37 | | | | | |
| <ul> <li>Mean MSK-HQ in Ortho hip and knee post-surgery = 42</li> </ul> | | | | | |
| MSK-HQ BL to 2Wk change score – Mean (SD) | | | | | |
| Percentage of patients who achieved MCID (>= 6 points) | | | | | |
| The Consumer Health Activation Index (CHAI) score – Mean (SD) <sup>a</sup> | | | | | |
| There is no reference value yet for this score | | | | | |
| Low (CHAI score 0-79) | | | | | |
| Moderate (CHAI score 80-94 | | | | | |
| High (CHAI score 95-100) | | | | | |
| The Consumer Health Activation Index (CHAI) BL-2W change | | | | | |
| score – Mean (SD) | | | | | |
| Percentage of patients who moved to an improved CHAI | | | | | |
| category | | | | | |
| Valuing Patients as Individuals Scale – Care and respect | | | | | |
| [scores range from 5 to 15: higher is better valued] | | | | | |
| The item asks if patients felt: | | | | | |
| - The clinic staff listened attentively to what they said | | | | | |
| - The clinic staff were very approachable and easy to talk to | | | | | |
| - The clinic staff treated me kindly | | | | | |
| There are no reference values yet, but this score is high | | | | | |
| Valuing Patients as Individuals – Understanding & engagement | | | | | |
| [scores range from 5 to 15: higher is better valued] | | | | | |
| The item asks if patients felt: | | | | | |
| - My problems were regarded as important by the therapist | | | | | |
| - The therapist answered all my questions | | | | | |
| - The therapist treated me as an intelligent human being | | | | | |
| There are no reference values yet, but this score is high | | | 1 | 1 | |

# Patient reported experience measures at 2 weeks

| Patient reported experience measures at 2 weeks |
|-------------------------------------------------------------|
| Friends and Family Test: |
| How likely are you to recommend this service to friends and |
| family if they need similar care or treatment? |
| Extremely likely |
| Likely |
| Neither likely nor unlikely |
| Unlikely |
| Extremely unlikely |
| Don't know |
| Was it easy for you to get to the clinic? |
| Very easy |
| Easy |
| Uncertain |
| Not easy |
| Not easy at all |
| Prefer not to say |
| Was the environment of the clinic okay? |

| Excellent environment |
|--------------------------------------------------------------------|
| Good environment |
| Uncertain |
| Poor environment |
| Very poor environment |
| Prefer not to say |
| As a result of your visit are you accessing less or more NHS care? |
| Much more care |
| More care |
| About the same care |
| Less care |
| Much less care |
| Prefer not to say |
| How much support was available to help you make decisions |
| about your treatment? |
| Excellent support |
| Good support |
| Uncertain |
| Poor support |
| Very poor support |
| Prefer not to say |
| How well do you feel you now know: a) Your treatment options? |
| Very well |
| Well |
| Uncertain |
| Not well |
| Not well at all |
| Prefer not to say |
| How well do you feel you now know: b) The pros and cons for |
| each option? |
| Very well |
| Well |
| Uncertain |
| Not well |
| Not well at all |
| Prefer not to say |

Three month follow up outcome measures

| Three month follow up outcome measures | Phase 1 | Phase 3 | Total | Mean (95% CI) | P-value |
|---|---|---|---|---|---|
| Global change in MSK condition since my clinic appointment | | | | | |
| (5 =much better to 1 = much worse- see below) – Mean (SD) | | | | | |
| Global change | | | | | |
| 5. Much better | | | | | |
| 4. Better | | | | | |
| 3. Same | | | | | |
| 2. Worse | | | | | |
| 1. Much worse | | | | | |
| Composite Scores | | | | | |
| Patient enablement index – Mean (SD) | | | | | |
| [score range is 0 to 12: higher scores = better empowerment] | | | | | |
| This items asks – "As a result of your visit to the clinic, do you | | | | | |
| feel you are:" (options - Much better=2, Better=1, Same=0) | | | | | |
| Able to understand your illness | | | | | |
| <ul> <li>Able to cope with your illness</li> </ul> | | | | | |
| Able to keep yourself healthy | | | | | |
| Able to cope with life | | | | | |
| <ul> <li>Confident about your health</li> </ul> | | | | | |
| Able to help yourself | | | | | |
| Reference values: | | | | | |
| In a GP sample patient mean PEI score was 4 points (1 wk later) | | | | | |
| MSK-HQ score – Mean (SD) | | | | | |
| Reference score at Follow-up: | | | | | |
| <ul> <li>Mean MSK-HQ in National FCP pilot = 41</li> </ul> | | | | | |
| <ul> <li>Mean MSK-HQ in Community physio = 42</li> </ul> | | | | | |
| <ul> <li>Mean MSK-HQ in GP sample = 37</li> </ul> | | | | | |
| Mean MSK-HQ in Ortho hip and knee post-surgery = 42 | | | | | |
| MSK-HQ BL to 3 month change score – Mean (SD) | | | | | |
| Percentage of patients who achieved MCID (>= 6 points) | | | | | |
| The Consumer Health Activation Index (CHAI) score – Mean (SD) <sup>a</sup> | | | | | |
| There is no reference value yet for this score | | | | | |
| The Consumer Health Activation Index (CHAI) BL-3M change | | | | _ | _ |
| score – Mean (SD) | | | | | |
| Low (CHAI score 0-79) | | | | | |
| Moderate (CHAI score 80-94 | | | | | |
| High (CHAI score 95-100) | | | | | |

#### Work measures

| WPAI Derived Measures: |
|---------------------------------------------------------------|
| Percent work time missed due to problem: |
| Percent impairment while working due to problem |
| Percent overall work impairment due to problem |
| Percent activity impairment due to problem |
| Work & Activity |
| Work status – Working |
| Hours missed from work in last 7 days because of problem- |
| Mean (SD) |
| Hours missed from work in last 7 days for other reasons- Mean |
| (SD) |
| Hours worked in last 7 days for other reasons - Mean (SD) |
| Joint and muscle symptoms affect your productivity while |
| working - Mean (SD) |
| Joint and muscle symptoms affect ability to do regular daily |
| activities, other than work - Mean (SD) |

#### **Patient Experience at 3 months**

| ratient Experience at 3 months | 1 | 1 |
|---|---|---|
| A | | |
| As a result of your visit are you accessing less or more NHS care? b [no baseline] | | |
| Much more care | | |
| More care | | |
| About the same care | | |
| Less care | | |
| Much less care | | |
| Prefer not to say | | |
| Patient thoughts about the MSK Tracker System | | |
| How useful did you find it? | | |
| Very useful | | |
| Useful | | |
| Uncertain | | |
| Not useful | | |
| Not useful at all | | |
| Prefer not to say | | |
| How easy was it to use? | | |
| Very easy | | |
| Easy | | |
| Uncertain | | |
| Not easy | | |
| Not easy at all | | |
| Prefer not to say | | |
| How well did it help you think about the issue related to the care for your joint and muscle symptoms? | | |
| Very well | | |
| Well | | |
| Uncertain | | |
| Not well | | |
| Not well at all | | |
| Prefer not to say | | |
| Did it increase any stress associated with your appointment? | | |
| Yes - increased stress a lot | | |
| Yes - increased stress a little | | |
| Made no difference | | |
| No - it reduced stress a little | | |
| No - it reduced stress a lot | | |

# 10. Appendices

# Figure 1 - Consort diagram



Figure 2 - Study Flow chart

